CLINICAL TRIAL: NCT02368704
Title: Role of Endoplasmic Reticulum Stress in the Pathophysiology of Type 2 Diabetes
Acronym: GLUCOSTRESS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: GLUCOSTRESS P 08 11 22
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2; Endoplasmic Reticulum Stress
Keywords: Endoplasmic Reticulum
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples. These samples will be anonymized, frozen and stored in the INSERM UMR-S 872 in the Cordeliers Research Center (Madame Fabienne Foufelle) under the responsibility of Professor Jean-François Gautier for a maximum period of 15 years, beyond which they will be destroyed. These samples will be destroyed at any time at the request of the patient. This DNA storage will be used to study genes related to the secretion of insulin and to identify other genes involved in the onset of diabetes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: control subjects with :
  * Nondiabetic subjects (blood glucose <7.0 mmol/l without hypoglycemic treatment).
  * The control subjects should be matched to patients for age (± 5 years), sex, and BMI (± 2 kg/m2).
  Interventions: Other: No intervention
- case: Diabetic patients with :
  * Having type 2 diabetes for at least 6 months
  * HbA1c ≤ 8%
  * Treat by lifestyle and dietary rules associated or not to a hypoglycemic therapy (metformin and / or sulfamid) and / or insulin secretors dependent glucose as inhibitors of DPP4 (dipeptidyl peptidase-4): Vildagliptin, Sitagliptin, Saxagliptin
  * No modification of hypoglycemic therapy and / or insulin secretors for at least 3 months
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to investigate whether Endoplasmic Reticulum (ER) stress pathway is activated in peripheral tissues (adipose tissue) in insulin resistant diabetic patients compared to healthy subjects normoglycemic matched for age and sex an to investigate whether ER stress pathway can be activated in response to insulin. Indeed, some preliminar on rates studies shows that ER stress pathway is activated by insulin in liver and adipose tissue showing that hyperinsulinemia might help trigger stress path ER.

For this, we propose a case control study of type 2 diabetic patients vs control subjects in which markers of ER stress will be evaluated from abdominal subcutaneous adipose tissue obtained before and after euglycemic hyperinsulinemic. We chose to consider adipose tissue subcutaneous rather than visceral adipose tissue for obvious reasons of lesser invasiveness.

ELIGIBILITY:
Inclusion Criteria:

* Specific criteria for diabetic patients:
* Having type 2 diabetes for at least 6 months
* HbA1c ≤ 8%
* Treated by lifestyle and dietary rules associated or not to a hypoglycemic therapy (metformin and / or sulfamid) and / or insulin secretors dependent glucose as inhibitors of DPP4 (dipeptidyl peptidase-4): Vildagliptin, Sitagliptin, Saxagliptin
* No modification of hypoglycemic therapy and / or insulin secretors for at least 3 months

Specific criteria for control subjects:

* Nondiabetic subjects (fasting blood glucose <7.0 mmol / l without hypoglycemic treatment).
* The control subjects should be matched to patients for age (± 5 years), sex, and BMI (± 2 kg/m2).

Common criteria for patients and control subjects:

* Aged 18 to 60 years
* Body Mass Index between 25 and 35 kg/m2
* Accepting the constraints of the protocol and who signed the informed consent
* Systolic blood pressure < 160 mmHg, diastolic blood pressure < 90 mm Hg (with or without antihypertensive treatment)
* Resting heart rate between 55 and 100 beats/min.
* Normal laboratory tests or not clinically significant abnormality for NFS platelets, PT, aPTT, fibrinogen ALT, AST, GGT, Serum electrolytes, urea, creatinine, Uric acid Triglycerides, total cholesterol, HDL cholesterol
* HCG negative blood (for female subjects)
* Affiliated to the Social Security.

Exclusion Criteria:

* Current infections or recent infections (<10 days)
* Neoplastic disorders (with the exception of carcinoma in situ of the cervix or cutaneous epithelioma), haematological, cardiovascular, psychiatric, neurological
* Poisoning smoking (>10 cigarettes per day, what ever the duration of intoxication)
* Treatment with insulin or glitazones Pregnancy, Breastfeeding
* Body Mass Index > 35 kg/m2
* Any drug taken for less than 8 days without the inclusion of minor analgesics (aspirin, paracetamol), anti-hypertensive medications, oral hypoglycemic (metformin and sulphonylureas) and insulin secretors dependent glucose as inhibitors of DPP4 (dipeptidyl peptidase-4) and oral contraceptives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with type 2 diabetes Healthy volunteers Adults
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Show an increase in markers of ER stress in fasting patients with type 2 diabetes | 2 days
  Protein expression markers of ER stress pathway BiP / GRP 78, CHOP, ATF4 EDEM and XBP-1

SECONDARY OUTCOMES:
Assess whether insulin induces an increase in markers of ER stress | 2 days
  Insulin sensitivity
Insulin secretion in response to glucose infusion | 2 days
Insulin secretion in response to arginine infusion | 2 days
Lipolysis on insulin | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, Paris, France